CLINICAL TRIAL: NCT01945710
Title: An Open-label, Multicenter, Multiple Dose, Phase 1 Study to Establish the Maximum Tolerated Dose of E7389 Liposomal Formulation in Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Limited (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E7389-E044-112; 2012-001184-69 (EudraCT Number)
Record Dates: First submitted 2013-09-16; First posted 2013-09-18 (Estimated); Results first posted 2019-07-23 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2018-03

CONDITIONS: Solid Tumors
Keywords: Tumors
MeSH Terms: conditions — Neoplasms | interventions — eribulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Eribulin-LF Schedule 1 (Experimental): Schedule 1: Eribulin-LF administered as IV infusion on Day 1 of a 21-day cycle starting at 1 mg/m^2 escalating up to 3.5 mg/m^2.
  Schedule 1a: Eribulin-LF administered as IV infusion on Day 1 of a 28-day cycle starting at 1 mg/m^2 escalating up to 3.5 mg/m^2 (only to be investigated in the event that a 21-day cycle is considered inappropriate).
  Interventions: Drug: Eribulin-LF
- Eribulin-LF Schedule 2 (Experimental): Schedule 2: Eribulin-LF administered as IV infusion on Day 1 and Day 15 of a 28-day cycle starting at 1 mg/m^2 escalating up to 3.5 mg/m^2 (only to be investigated in the event that a 21-day cycle is considered appropriate).
  Interventions: Drug: Eribulin-LF

INTERVENTIONS:
Drug: Eribulin-LF
  Other Names: E7389-liposomal formulation (E7389-LF); Eribulin mesylate; Eribulin mesilate

SUMMARY:
Study E7389-E044-112 is a Phase 1 study designed to assess the safety, tolerability and preliminary efficacy of eribulin-liposomal formulation (E7389-LF) in patients with solid tumors. This dose-escalation study will determine the maximum tolerated dose, dosing schedules tested, the dose schedule regimen with a more favorable tolerability profile, and a preliminary indication of efficacy.

DETAILED DESCRIPTION:
This is a Phase 1 first-in-human, non-randomized (individuals will not be assigned by chance to study treatments), open-label (individuals will know the identity of study treatments), multicenter, 2-part, dose-escalation study to evaluate the safety, pharmacokinetics (study of what the body does to a drug) of eribulin-LF administered intravenously to patients with solid tumors. Each treatment cycle will be 21 days (Schedule 1) or 28 days (Schedule 1a or 2). Part 1 is the dose-escalation phase, which will be guided by pharmacokinetics and safety. Three to 6 new patients will be enrolled in sequential cohorts (first cohort will receive the starting dose and subsequent cohorts will receive increased doses of eribulin-LF). Enrollment in each cohort will be staggered; the second and third participant in every cohort will not be dosed until the first patient in that cohort completes 2 weeks of Cycle 1. If no dose-limiting toxicities (DLTs) have been observed during the first 2 week of Cycle 1 in the first patient, the second and third patients in the cohort will initiate treatment. Enrollment will be first initiated into cohort 1 of Schedule 1 (dosing on Day 1 of 21 day cycle). Interim analysis will be conducted upon completion of this cohort. The following decisions will be made based upon the results of the interim analysis 1) proceed with escalating to next dose level (cohort 2) of Schedule 1 (dosing on Day 1 of 21 day cycle) and initiate cohort 1 of Schedule 2 (dosing on Day 1 and Day 15 of 28 day cycle), or 2) discontinue plans to evaluate Schedule 2 and initiate Schedule 1a (dosing on Day 1 of 28 day cycle).

After the last patient in each cohort completes Cycle 1, the safety for DLT determination will be evaluated and a decision will be made on whether to escalate the dose in a new cohort of 3 to 6 new patients. Dose escalation will halt when the maximum tolerated dose (MTD) is reached. The total number of patients to be enrolled in Part 1 will depend on the dose level at which the DLT will be achieved. After MTD for each schedule is determined, patients will be enrolled into Expansion Part of the study to confirm safety and tolerability of each dosing schedule. Nine to 12 patients will be treated with MTD for each schedule for 6 cycles. The total study duration for each participant will be approximately 18 months.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older.
2. Histological or cytological evidence of an unresectable or refractory solid tumor.
3. Participants who have at least one measurable lesion (long axis in non-lymph node: greater than or equal to 10 millimeters (mm); short axis in lymph node: greater than or equal to 15 mm) based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 in the Expansion Part.
4. Adequate liver function as evidenced by bilirubin less than or equal to 1.5 times the upper limits of normal (ULN) and alkaline phosphatase (ALP), alanine aminotransferase (ALT), and aspartate aminotransferase (AST) less than or equal to 3 x ULN (in the case of liver metastases less than or equal to 5 x ULN). In case ALP is greater than 3 x ULN (in absence of liver metastases) or greater than 5 x ULN (in presence of liver metastases) AND participant also is known to have bone metastases, the liver specific ALP must be separated from the total and used to assess the liver function instead of the total ALP.
5. Adequate renal function as evidenced by serum creatinine less than or equal to 2.0 milligrams/deciliter (mg/dL) (177 micromole/liter (umol/L)) or calculated creatinine clearance greater than or equal to 40 milliliter/minute (mL/min) per the Cockcroft and Gault formula.
6. Adequate bone marrow function as evidenced by absolute neutrophil count (ANC) greater than or equal to 1.5 x 10^9/liter (L), hemoglobin greater than or equal to 9 grams/deciliter (g/dL) (5.5 millimol/liter (mmol/L)) and platelet count greater than or equal to 100 x 10^9/L.
7. Females must not be lactating or pregnant at Screening or Baseline (as documented by a negative beta-human chorionic gonadotropin [B-hCG]). A separate baseline assessment is required if a negative screening pregnancy test was obtained more than 72 hours before the first dose of study drug.
8. All females will be considered to be of childbearing potential unless they are postmenopausal (amenorrheic for at least 12 consecutive months, in the appropriate age group and without other known or suspected cause) or have been sterilized surgically (i.e., bilateral tubal ligation, total hysterectomy or bilateral oophorectomy, all with surgery at least one month before dosing).
9. Females of childbearing potential must not have had unprotected sexual intercourse within 30 days before study entry and must agree to use two highly effective methods of contraception (e.g., total abstinence, an intrauterine device, a double-barrier method [condom and occlusive cap - diaphragm or cervical/vault caps - with spermicidal foam/gel/film/cream/suppository], a contraceptive implant, an oral contraceptive, or have a vasectomized partner with confirmed azoospermia) throughout the entire study period and for 30 days after study drug discontinuation. If currently abstinent, the participant must agree to use a double barrier method with spermicide as described above if she becomes sexually active during the study period or for 30 days after study drug discontinuation. Females who are using hormonal contraceptives must have been on a stable dose of the same hormonal contraceptive product for at least 4 weeks before dosing and must continue to use the same contraceptive during the study and for 30 days after study drug discontinuation.
10. Male participants must have had a successful vasectomy (confirmed azoospermia) or they and their female partners must meet the criteria above (i.e., not of childbearing potential or practicing highly effective contraception throughout the study period and for 30 days after study drug discontinuation). No sperm donation is allowed during the study period and for 30 days after study drug discontinuation.
11. Provide written informed consent.
12. Willing and able to comply with all aspects of the protocol.

Exclusion Criteria:

1. Females who are pregnant (positive B-hCG [or hCG] test) or breastfeeding.
2. Participants who have received any anticancer therapy within 21 days prior to study entry for cytotoxic agents (42 days for mitomycin C and nitrosoureas), radiotherapy, hormonal, biological (including humanized antibodies) and targeted agents, or within 30 days for an investigational agent.
3. Participants who have not recovered from acute toxicities as a result of prior anti-cancer therapy to less than Grade 2, according to Common Terminology Criteria for Adverse Events (CTCAE), except alopecia.
4. Participants who have previously been treated with eribulin-LF.
5. Radiation therapy encompassing greater than 30% of the bone marrow.
6. Major surgery within 21 days prior to enrollment.
7. Pre-existing peripheral neuropathy greater than CTCAE Grade 1.
8. Significant cardiovascular impairment, defined as:

   1. Congestive heart failure greater than Class II according to the New York Heart Association.
   2. Unstable angina or myocardial infarction within 6 months of enrollment, or cardiac arrhythmia requiring treatment.
   3. A clinically significant electrocardiogram (ECG) abnormality, including a marked baseline prolonged QT/QTc interval (e.g., a repeated demonstration of a QTc interval greater than 500 milliseconds (ms)).
   4. A history of risk factors for torsade de pointes (e.g., heart failure, hypokalemia, family history of long QT Syndrome) or the use of concomitant medications that prolonged the QT/QTc interval.
9. Evidence of clinically significant disease (e.g., cardiac, respiratory, gastrointestinal, renal disease) that in the opinion of the investigator(s) could affect the participant's safety or interfere with the study assessments.
10. Diagnosed with meningeal carcinomatosis.
11. Participants with brain or subdural metastases are not eligible, unless they have completed local therapy and have discontinued the use of corticosteroids for this indication for at least 4 weeks prior to enrollment. Any symptom(s) attributed to brain metastases must be stable for at least 4 weeks prior to enrollment, and radiographic stability should be confirmed by comparing a brain scan (CT with contrast or MRI with and without contrast) performed during the Screening Period to a brain scan performed at least 4 weeks earlier using the same modality.
12. Any serious concomitant illness or infection requiring treatment: known active human immunodeficiency virus (HIV) infection, hepatitis B, or hepatitis C infection (asymptomatic positive serology is not exclusionary).
13. Pulmonary lymphangitic involvement that results in pulmonary dysfunction requiring active treatment, including the use of oxygen.
14. History of drug or alcohol dependency or abuse within approximately the last 2 years or current use of illegal recreational drugs.
15. Known intolerance to Halaven (eribulin-LF; E7389-LF) or any of the excipients.
16. Any medical or other condition that in the opinion of the investigator(s) would preclude the participant's participation in a clinical study.
17. Scheduled for surgery during the study.
18. Participants with body mass index (BMI) less than 35.
19. Participants with proven abdominal malignancy with concurrent refractory ascites defined by one of the following criteria:

    1. Symptomatic ascites (more than 2 L) that did not respond clinically to at least 2 weeks of diuretics OR
    2. Removal of at least 10 L in the preceding 2 months for symptoms relief OR
    3. Symptomatic ascites that recurred on at least three occasions within a 2 month period despite diuretic treatment.
20. Participants with concurrent refractory pleural effusion defined by the following criteria:

    1. Symptomatic pleural effusion that did not respond clinically to the treatment and needed pleural drainage in the preceding 2 months for symptoms relief OR
    2. Recurrent symptomatic pleural effusion on at least three occasions within a 2 month period despite treatment.
21. Currently enrolled in another clinical trial or used any investigational drug or device within 30 days or 5X the half-life, whichever is longer preceding informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2012-12-11 (Actual); Primary Completion 2015-10 (Actual); Study Completion 2016-05-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United Kingdom (4):
  - Royal Marsden Hospital, Sutton, Surrey
  - Beatson West of Scotland Cancer Centre, Glasgow
  - UCL Cancer Institute, London
  - The Christie NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Eisai's data sharing commitment and further information on how to request data can be found on our website http://eisaiclinicaltrials.com/.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Total 71 subjects were screened for entry into the study of which 62 were enrolled and 9 were screen failures. Of the 9 screen failures, 7 did not meet the inclusion/exclusion criteria, 1 experienced an adverse event that led to screening discontinuation, and 1 did not proceed to treatment in the study. Of the 62 enrolled, 58 subjects were treated.
Groups:
- Schedule 1 Dose Escalation Cohort: 1.0 mg/m^2 Eribulin-LF: Dose Escalation Cohort: Eribulin-LF (1.0 milligram per square meter [mg/m^2]) was administered as an IV infusion on Day 1 of a 21-day cycle starting at 1 mg/m^2 escalating until intolerable toxicity, disease progression or death.
- Schedule 1 Dose Escalation Cohort: 1.4 mg/m^2 Eribulin-LF: Dose Escalation Cohort: Eribulin-LF (1.4 mg/m^2) was administered as an IV infusion on Day 1 of a 21-day cycle starting at 1 mg/m^2 escalating until intolerable toxicity, disease progression or death.
- Schedule 1 Dose Escalation Cohort: 1.5 mg/m^2 Eribulin-LF: Dose Escalation Cohort: Eribulin-LF (1.5 mg/m^2) was administered as an IV infusion on Day 1 of a 21-day cycle starting at 1 mg/m^2 escalating until intolerable toxicity, disease progression or death.
- Schedule 2 Dose Escalation Cohort: 1.0 mg/m^2 Eribulin-LF: Dose Escalation Cohort: Eribulin-LF (1.0 mg/m^2) was administered as an IV infusion on Day 1 and Day 15 of a 28-day cycle starting at 1 mg/m^2 escalating until intolerable toxicity, disease progression or death.
- Schedule 2 Dose Escalation Cohort: 1.5 mg/m^2 Eribulin-LF: Dose Escalation Cohort: Eribulin-LF (1.5 mg/m^2) was administered as an IV infusion on Day 1 and Day 15 of a 28-day cycle starting at 1 mg/m^2 escalating until intolerable toxicity, disease progression or death.
- Schedule 2 Dose Escalation Cohort: 2.0 mg/m^2 Eribulin-LF: Dose Escalation Cohort: Eribulin-LF (2.0 mg/m^2) was administered as an IV infusion on Day 1 and Day 15 of a 28-day cycle starting at 1 mg/m^2 escalating until intolerable toxicity, disease progression or death.
- Schedule 2 Expansion Cohort: 1.5 mg/m^2 Eribulin-LF: Dose Expansion Cohort: Eribulin-LF (1.5 mg/m^2) was administered as an IV infusion on Day 1 and Day 15 of a 28-day cycle.
Period: Overall Study
Arm/Group | Schedule 1 Dose Escalation Cohort: 1.0 mg/m^2 Eribulin-LF | Schedule 1 Dose Escalation Cohort: 1.4 mg/m^2 Eribulin-LF | Schedule 1 Dose Escalation Cohort: 1.5 mg/m^2 Eribulin-LF | Schedule 2 Dose Escalation Cohort: 1.0 mg/m^2 Eribulin-LF | Schedule 2 Dose Escalation Cohort: 1.5 mg/m^2 Eribulin-LF | Schedule 2 Dose Escalation Cohort: 2.0 mg/m^2 Eribulin-LF | Schedule 2 Expansion Cohort: 1.5 mg/m^2 Eribulin-LF
Started | 7 | 6 | 7 | 3 | 9 | 3 | 23
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 7 | 6 | 7 | 3 | 9 | 3 | 23
Not completed — Progressive Disease | 5 | 4 | 3 | 2 | 7 | 3 | 19
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 2 | 0 | 3 | 1 | 1 | 0 | 4
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set (SAS) was the group of participants who received study drug and had at least 1 post-dose safety assessment.
Groups:
- Schedule 1 Dose Escalation Cohort: 1.0 mg/m^2 Eribulin-LF: Dose Escalation Cohort: Eribulin-LF (1.0 mg/m^2) was administered as an IV infusion on Day 1 of a 21-day cycle starting at 1 mg/m^2 escalating until intolerable toxicity, disease progression or death.
- Total: Total of all reporting groups
Arm/Group | Schedule 1 Dose Escalation Cohort: 1.0 mg/m^2 Eribulin-LF | Schedule 1 Dose Escalation Cohort: 1.4 mg/m^2 Eribulin-LF | Schedule 1 Dose Escalation Cohort: 1.5 mg/m^2 Eribulin-LF | Schedule 2 Dose Escalation Cohort: 1.0 mg/m^2 Eribulin-LF | Schedule 2 Dose Escalation Cohort: 1.5 mg/m^2 Eribulin-LF | Schedule 2 Dose Escalation Cohort: 2.0 mg/m^2 Eribulin-LF | Schedule 2 Expansion Cohort: 1.5 mg/m^2 Eribulin-LF | Total
Number analyzed (Participants) | 7 | 6 | 7 | 3 | 9 | 3 | 23 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.3 (9.57) | 54.2 (12.22) | 59.0 (12.26) | 65.3 (2.08) | 62.9 (6.13) | 59.0 (16.52) | 56.0 (9.31) | 58.6 (9.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 3 | 1 | 4 | 1 | 23 | 38
  Male | 3 | 4 | 4 | 2 | 5 | 2 | 0 | 20

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Eribulin-LF
Description: The MTD was defined as the highest dose level at which no more than 1/6 participants experienced a dose limiting toxicity (DLTs), with the next higher dose having at least 2 of 3 or 2 of 6 participants experiencing DLTs. MTD was determined by summarizing the number and percentage of participants with DLTs for the first cycle, by study dosing schedule, initial dosing level and overall for the dose escalation part. For participants who continued to Cycle 2, the DLTs which occurred from 1st dose up to the day before Day 1 of Cycle 2 were counted. For participants who discontinued before Cycle 2, the DLTs which occurred from 1st dose up to Day 21 (Schedule 1) or Day 28 (Schedule 2) of Cycle 1 were counted. DLTs were evaluated and graded based on the National Cancer Institutes (NCI)'s Common Terminology Criteria for Adverse Events (CTCAE) version 4.03.
Time Frame: Schedule 1: Cycle 1 (21 days); Schedule 2: Cycle 1 (28 days)
Population: Dose finding analysis set is all participants in the dose escalation part who completed Cycle 1 treatment and were evaluated for DLTs, and those who discontinued during Cycle 1 due to DLT.
Measure: Number; unit: mg/m^2
Groups:
- Schedule 1: Total Escalation Cohorts: Eribulin-LF (1.0 mg/m^2, 1.4 mg/m^2, or 1.5 mg/m^2) was administered as an IV infusion on Day 1 of a 21-day cycle starting at 1 mg/m^2 escalating until intolerable toxicity, disease progression or death.
- Schedule 2: Total Dose Escalation and Expansion: Dose Escalation Cohort: Eribulin-LF (1.0 mg/m^2, 1.5 mg/m^2, or 2.0 mg/m^2) was administered as an IV infusion on Day 1 and Day 15 of a 28-day cycle starting at 1 mg/m^2 escalating until intolerable toxicity, disease progression or death.
  Expansion Cohort: Eribulin-LF (1.5 mg/m^2) was administered as an IV infusion on Day 1 and Day 15 of a 28-day cycle.
Arm/Group | Schedule 1: Total Escalation Cohorts | Schedule 2: Total Dose Escalation and Expansion
Number analyzed (Participants) | 18 | 12
mg/m^2 | 1.4 | 1.5

2. Primary Outcome: Dose Limiting Toxicities at the Indicated Dose Levels, as an Assessment of Dosing Frequency
Description: DLTs were evaluated for both Schedule 1 and Schedule 2. DLTs were defined as neutropenia grade 4 that lasted more than 5 days, neutropenia grade 3 or 4 complicated by fever and/or infection (absolute neutrophil count (ANC) less than 1.0 x 10^9/liter, fever greater than or equal to 38.5 degrees Celsius), thrombocytopenia grade 4 of any duration, thrombocytopenia grade 3 complicated by bleeding and/or requiring platelet or blood transfusion, hypersensitivity reaction grade 3 or 4 including allergy reactions or anaphylaxis; symptomatic bronchospasm requiring parenteral medication(s) with our without urticarial; allergy-related edema/angioedema, or other grade 3 or 4 clinically significant non-hematologic toxicities (except for inadequately treated nausea and /or vomiting) considered related to study drug. Participants with two or more adverse events in the same system organ class (or with the same preferred term) was counted only once for that system organ class (or preferred term).
Time Frame: Cycle 1 of Dose Escalation part in Schedule 1 and Schedule 2
Population: Dose-finding analysis set included all participants in the dose escalation part who completed Cycle 1 treatment and were evaluated for DLTs and those who discontinued during Cycle 1 due to DLTs.
Measure: Count of Participants; unit: Participants
Arm/Group | Schedule 1 Dose Escalation Cohort: 1.0 mg/m^2 Eribulin-LF | Schedule 1 Dose Escalation Cohort: 1.4 mg/m^2 Eribulin-LF | Schedule 1 Dose Escalation Cohort: 1.5 mg/m^2 Eribulin-LF | Schedule 2 Dose Escalation Cohort: 1.0 mg/m^2 Eribulin-LF | Schedule 2 Dose Escalation Cohort: 1.5 mg/m^2 Eribulin-LF | Schedule 2 Dose Escalation Cohort: 2.0 mg/m^2 Eribulin-LF
Number analyzed (Participants) | 6 | 6 | 6 | 3 | 6 | 3
Participants
  Transaminases increased | 0 | 0 | 1 | 0 | 0 | 0
  Hypophosphataemia | 0 | 0 | 1 | 0 | 0 | 0
  Febrile neutropenia | 0 | 0 | 0 | 0 | 1 | 0
  Neutropenia | 0 | 0 | 0 | 0 | 0 | 1
  Stomatitis | 0 | 0 | 0 | 0 | 1 | 0
  Alanine aminotransferase increased | 0 | 0 | 0 | 0 | 0 | 1

3. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) as a Measure of Safety and Tolerability of Eribulin-LF
Description: Safety was assessed by the monitoring and recording of all adverse events (AEs), and serious AEs (SAEs), regular monitoring of hematology, clinical chemistry, and urine values; periodic measurement of vital signs, electrocardiograms; and the performance of physical examinations. For each row category, a participant with two or more adverse events in that category is counted only once. Treatment-related TEAEs include TEAEs that were considered by the Investigator to be possibly or probably related to study drug and TEAEs with a missing relationship to study drug.
Time Frame: From date of first dose until 30 days after the final dose of study drug, up to approximately 3 years 6 months
Population: The SAS was the group of participants who received study drug and had at least 1 post-dose safety assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Schedule 1 Dose Escalation Cohort: 1.0 mg/m^2 Eribulin-LF | Schedule 1 Dose Escalation Cohort: 1.4 mg/m^2 Eribulin-LF | Schedule 1 Dose Escalation Cohort: 1.5 mg/m^2 Eribulin-LF | Schedule 2 Dose Escalation Cohort: 1.0 mg/m^2 Eribulin-LF | Schedule 2 Dose Escalation Cohort: 1.5 mg/m^2 Eribulin-LF | Schedule 2 Dose Escalation Cohort: 2.0 mg/m^2 Eribulin-LF | Schedule 2 Expansion Cohort: 1.5 mg/m^2 Eribulin-LF
Number analyzed (Participants) | 7 | 6 | 7 | 3 | 9 | 3 | 23
Participants
  TEAEs | 7 | 6 | 7 | 3 | 9 | 3 | 23
  Treatment-related TEAEs | 6 | 6 | 6 | 3 | 6 | 3 | 22
  Serious TEAEs | 1 | 2 | 6 | 1 | 3 | 2 | 9
  TEAEs leading to drug dose adjustment | 3 | 2 | 3 | 1 | 3 | 3 | 17
  TEAEs leading to drug withdrawal | 1 | 0 | 2 | 0 | 0 | 0 | 2
  TEAEs leading to dose reduction | 0 | 0 | 1 | 0 | 1 | 2 | 0
  TEAEs leading to dose interruption | 2 | 2 | 1 | 1 | 3 | 3 | 16

4. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Eribulin-LF
Description: Blood samples for Schedule 1 were drawn on Cycle 1/Day 1 and Cycle 3/Day 1 predose, 15 minutes (min) after the start of infusion (SOI), 5 min after the end of infusion (EOI), 0.5, 1, 2, 4, 6, 8, and 24 hours (h) postdose, and Day 4, Day 7, Day 9, and Day 11. Blood samples for Schedule 2 were drawn on Cycle 1/Day 1 and Day 15 and Cycle 3/Day 1 and Day 15 predose, 15 min after the SOI, 5 min after the EOI, 0.5, 1, 2, 4, 6, 8, and 24 h postdose, and Day 4, Day 7, Day 9 and Day 11. Some participants followed a different pharmacokinetic (PK) assessment schedule prior to protocol amendment 3. Plasma concentrations of eribulin-LF were determined using a validated liquid chromatography-tandem mass spectrometry (LC/MS/MS) method. Plasma PK data were analyzed using a noncompartmental analysis approach to obtain individual participant estimates of Cmax, which was then summarized as the mean and standard deviation for all participants and expressed as nanograms/milliliter (ng/mL).
Time Frame: Schedule 1: Cycle 1/Day 1 and Cycle 3/Day 1; Schedule 2: Cycle 1/Day 1 and Day 15 and Cycle 3/Day 1 and Day 15
Population: The PK analysis set was the group of participants who had sufficient PK data to derive at least one PK parameter.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Schedule 1 Dose Escalation Cohort: 1.0 mg/m^2 Eribulin-LF | Schedule 1 Dose Escalation Cohort: 1.4 mg/m^2 Eribulin-LF | Schedule 1 Dose Escalation Cohort: 1.5 mg/m^2 Eribulin-LF | Schedule 2 Dose Escalation Cohort: 1.0 mg/m^2 Eribulin-LF | Schedule 2 Dose Escalation Cohort: 1.5 mg/m^2 Eribulin-LF | Schedule 2 Dose Escalation Cohort: 2.0 mg/m^2 Eribulin-LF
Number analyzed (Participants) | 6 | 6 | 7 | 3 | 9 | 3
ng/mL | 1986.2 (3084.77) | 1119.8 (205.71) | 1211.3 (293.35) | 665.3 (125.13) | 1213.3 (259.42) | 1473.3 (47.26)

5. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) of Eribulin-LF
Description: Blood samples for Schedule 1 were drawn on Cycle 1/Day 1 and Cycle 3/Day 1 predose, 15 min after the SOI, 5 min after the EOI, 0.5, 1, 2, 4, 6, 8, and 24 h postdose, and Day 4, Day 7, Day 9, and Day 11. Blood samples for Schedule 2 were drawn on Cycle 1/Day 1 and Day 15 and Cycle 3/Day 1 and Day 15 predose, 15 min after the SOI, 5 min after the EOI, 0.5, 1, 2, 4, 6, 8, and 24 h postdose, and Day 4, Day 7, Day 9 and Day 11. Some participants followed a different PK assessment schedule prior to protocol amendment 3. Plasma concentrations of eribulin-LF were determined using a validated LC/MS/MS method. Plasma PK data were analyzed using a noncompartmental analysis approach to obtain individual participant estimates of Tmax, which was then summarized as the median and full range for all participants and expressed as hours.
Time Frame: Schedule 1: Cycle 1/Day 1 and Cycle 3/Day 1; Schedule 2: Cycle 1/Day 1 and Day 15 and Cycle 3/Day 1 and Day 15
Population: The PK analysis set was the group of participants who had sufficient PK data to derive at least one PK parameter.
Measure: Median (Full Range); unit: hours
Arm/Group | Schedule 1 Dose Escalation Cohort: 1.0 mg/m^2 Eribulin-LF | Schedule 1 Dose Escalation Cohort: 1.4 mg/m^2 Eribulin-LF | Schedule 1 Dose Escalation Cohort: 1.5 mg/m^2 Eribulin-LF | Schedule 2 Dose Escalation Cohort: 1.0 mg/m^2 Eribulin-LF | Schedule 2 Dose Escalation Cohort: 1.5 mg/m^2 Eribulin-LF | Schedule 2 Dose Escalation Cohort: 2.0 mg/m^2 Eribulin-LF
Number analyzed (Participants) | 6 | 6 | 7 | 3 | 9 | 3
hours | 1.95 [0.92 to 4.77] | 2.835 [1.50 to 5.00] | 2.00 [0.98 to 5.08] | 0.82 [0.23 to 0.95] | 1.13 [0.95 to 2.92] | 2.10 [1.18 to 2.17]

6. Secondary Outcome: Plasma Half-life (t1/2) of Eribulin-LF
Description: Blood samples for Schedule 1 were drawn on Cycle 1/Day 1 and Cycle 3/Day 1 predose, 15 min after SOI, 5 min after EOI, 0.5, 1, 2, 4, 6, 8, and 24 h postdose, and Day 4, Day 7, Day 9, and Day 11. Blood samples for Schedule 2 were drawn on Cycle 1/Day 1 and Day 15 and Cycle 3/Day 1 and Day 15 predose, 15 min after the SOI, 5 min after the EOI, 0.5, 1, 2, 4, 6, 8, and 24 h postdose, and Day 4, Day 7, Day 9 and Day 11. Plasma concentrations of eribulin-LF were determined using a validated LC/MS/MS method. Plasma PK data were analyzed using a noncompartmental analysis approach to obtain individual participant estimates of t1/2, which was then summarized as the mean and standard deviation for all participants and expressed in hours.
Time Frame: Schedule 1: Cycle 1/Day 1 and Cycle 3/Day 1; Schedule 2: Cycle 1/Day 1 and Day 15 and Cycle 3/Day 1 and Day 15
Population: The PK analysis set was the group of participants who had sufficient PK data to derive at least one PK parameter.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Schedule 1 Dose Escalation Cohort: 1.0 mg/m^2 Eribulin-LF | Schedule 1 Dose Escalation Cohort: 1.4 mg/m^2 Eribulin-LF | Schedule 1 Dose Escalation Cohort: 1.5 mg/m^2 Eribulin-LF | Schedule 2 Dose Escalation Cohort: 1.0 mg/m^2 Eribulin-LF | Schedule 2 Dose Escalation Cohort: 1.5 mg/m^2 Eribulin-LF | Schedule 2 Dose Escalation Cohort: 2.0 mg/m^2 Eribulin-LF
Number analyzed (Participants) | 6 | 6 | 7 | 3 | 9 | 3
hours | 22.20 (2.212) | 23.62 (4.614) | 34.87 (19.374) | 36.83 (32.679) | 28.07 (9.386) | 21.13 (3.837)

7. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time 0 Time of Last Quantifiable Concentration (AUC(0-t) ) of Eribulin-LF
Description: Blood samples for Schedule 1 were drawn on Cycle 1/Day 1 and Cycle 3/Day 1 predose, 15 min after SOI, 5 min after EOI, 0.5, 1, 2, 4, 6, 8, and 24 h postdose, and Day 4, Day 7, Day 9, and Day 11. Blood samples for Schedule 2 were drawn on Cycle 1/Day 1 and Day 15 and Cycle 3/Day 1 and Day 15 predose, 15 min after the SOI, 5 min after the EOI, 0.5, 1, 2, 4, 6, 8, and 24 h postdose, and Day 4, Day 7, Day 9 and Day 11. Plasma concentrations of eribulin-LF were determined using a validated LC/MS/MS method. Plasma PK data were analyzed using a noncompartmental analysis approach to obtain individual participant estimates of AUC(0-t), which was then summarized as the mean and standard deviation for all participants and expressed in nanograms*hour/milliliter (ng*hr/mL).
Time Frame: Schedule 1: Cycle 1/Day 1 and Cycle 3/Day 1; Schedule 2: Cycle 1/Day 1 and Day 15 and Cycle 3/Day 1 and Day 15
Population: The PK analysis set was the group of participants who had sufficient PK data to derive at least one PK parameter.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Schedule 1 Dose Escalation Cohort: 1.0 mg/m^2 Eribulin-LF | Schedule 1 Dose Escalation Cohort: 1.4 mg/m^2 Eribulin-LF | Schedule 1 Dose Escalation Cohort: 1.5 mg/m^2 Eribulin-LF | Schedule 2 Dose Escalation Cohort: 1.0 mg/m^2 Eribulin-LF | Schedule 2 Dose Escalation Cohort: 1.5 mg/m^2 Eribulin-LF | Schedule 2 Dose Escalation Cohort: 2.0 mg/m^2 Eribulin-LF
Number analyzed (Participants) | 6 | 6 | 7 | 3 | 9 | 3
ng*h/mL | 27016.7 (5022.91) | 30333.3 (6068.83) | 33457.1 (13808.68) | 12763.3 (7917.72) | 32201.1 (11854.28) | 49066.7 (7605.48)

8. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time 0 to Infinity (AUC(0-inf)) of Eribulin-LF
Description: Blood samples for Schedule 1 were drawn on Cycle 1/Day 1 and Cycle 3/Day 1 predose, 15 min after SOI, 5 min after EOI, 0.5, 1, 2, 4, 6, 8, and 24 h postdose, and Day 4, Day 7, Day 9, and Day 11. Blood samples for Schedule 2 were drawn on Cycle 1/Day 1 and Day 15 and Cycle 3/Day 1 and Day 15 predose, 15 min after the SOI, 5 min after the EOI, 0.5, 1, 2, 4, 6, 8, and 24 h postdose, and Day 4, Day 7, Day 9 and Day 11. Plasma concentrations of eribulin-LF were determined using a validated LC/MS/MS method. Plasma PK data were analyzed using a noncompartmental analysis approach to obtain individual participant estimates of AUC(0-inf), which was then summarized as the mean and standard deviation for all participants and expressed in ng*hr/mL.
Time Frame: Schedule 1: Cycle 1/Day 1 and Cycle 3/Day 1; Schedule 2: Cycle 1/Day 1 and Day 15 and Cycle 3/Day 1 and Day 15
Population: The PK analysis set was the group of participants who had sufficient PK data to derive at least one PK parameter.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Schedule 1 Dose Escalation Cohort: 1.0 mg/m^2 Eribulin-LF | Schedule 1 Dose Escalation Cohort: 1.4 mg/m^2 Eribulin-LF | Schedule 1 Dose Escalation Cohort: 1.5 mg/m^2 Eribulin-LF | Schedule 2 Dose Escalation Cohort: 1.0 mg/m^2 Eribulin-LF | Schedule 2 Dose Escalation Cohort: 1.5 mg/m^2 Eribulin-LF | Schedule 2 Dose Escalation Cohort: 2.0 mg/m^2 Eribulin-LF
Number analyzed (Participants) | 6 | 6 | 7 | 3 | 9 | 3
ng*h/mL | 27283.3 (5087.80) | 30366.7 (6062.23) | 33614.3 (13874.13) | 12820.0 (7870.43) | 32364.4 (11900.94) | 49400.0 (8179.85)

9. Secondary Outcome: Total Body Clearance (CL) of Eribulin-LF
Description: Blood samples for Schedule 1 were drawn on Cycle 1/Day 1 and Cycle 3/Day 1 predose, 15 min after the SOI, 5 min after the EOI, 0.5, 1, 2, 4, 6, 8, and 24 h postdose, and Day 4, Day 7, Day 9, and Day 11. Blood samples for Schedule 2 were drawn on Cycle 1/Day 1 and Day 15 and Cycle 3/Day 1 and Day 15 predose, 15 min after the SOI, 5 min after the EOI, 0.5, 1, 2, 4, 6, 8, and 24 h postdose, and Day 4, Day 7, Day 9 and Day 11. Some participants followed a different PK assessment schedule prior to protocol amendment 3. Plasma concentrations of eribulin-LF were determined using a validated LC/MS/MS method. Plasma PK data were analyzed using a noncompartmental analysis approach to obtain individual participant estimates of CL, which was then summarized as the mean and standard deviation for all participants and expressed as milliliter/hour (mL/h).
Time Frame: Schedule 1: Cycle 1/Day 1 and Cycle 3/Day 1; Schedule 2: Cycle 1/Day 1 and Day 15 and Cycle 3/Day 1 and Day 15
Population: The PK analysis set was the group of participants who had sufficient PK data to derive at least one PK parameter.
Measure: Mean (Standard Deviation); unit: mL/h
Arm/Group | Schedule 1 Dose Escalation Cohort: 1.0 mg/m^2 Eribulin-LF | Schedule 1 Dose Escalation Cohort: 1.4 mg/m^2 Eribulin-LF | Schedule 1 Dose Escalation Cohort: 1.5 mg/m^2 Eribulin-LF | Schedule 2 Dose Escalation Cohort: 1.0 mg/m^2 Eribulin-LF | Schedule 2 Dose Escalation Cohort: 1.5 mg/m^2 Eribulin-LF | Schedule 2 Dose Escalation Cohort: 2.0 mg/m^2 Eribulin-LF
Number analyzed (Participants) | 6 | 6 | 7 | 3 | 9 | 3
mL/h | 60.15 (17.500) | 75.93 (22.818) | 80.90 (29.390) | 148.63 (61.905) | 95.82 (58.289) | 65.37 (8.465)

10. Secondary Outcome: Volume of Distribution (Vd) of Eribulin-LF
Description: Blood samples for Schedule 1 were drawn on Cycle 1/Day 1 and Cycle 3/Day 1 predose, 15 min after the SOI, 5 min after the EOI, 0.5, 1, 2, 4, 6, 8, and 24 h postdose, and Day 4, Day 7, Day 9, and Day 11. Blood samples for Schedule 2 were drawn on Cycle 1/Day 1 and Day 15 and Cycle 3/Day 1 and Day 15 predose, 15 min after the SOI, 5 min after the EOI, 0.5, 1, 2, 4, 6, 8, and 24 h postdose, and Day 4, Day 7, Day 9 and Day 11. Some participants followed a different PK assessment schedule prior to protocol amendment 3. Plasma concentrations of eribulin-LF were determined using a validated LC/MS/MS method. Plasma PK data were analyzed using a noncompartmental analysis approach to obtain individual participant estimates of Vd, which was then summarized as the mean and standard deviation for all participants and expressed as milliliters (mL).
Time Frame: Schedule 1: Cycle 1/Day 1 and Cycle 3/Day 1; Schedule 2: Cycle 1/Day 1 and Day 15 and Cycle 3/Day 1 and Day 15
Population: The PK analysis set was the group of participants who had sufficient PK data to derive at least one PK parameter.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Schedule 1 Dose Escalation Cohort: 1.0 mg/m^2 Eribulin-LF | Schedule 1 Dose Escalation Cohort: 1.4 mg/m^2 Eribulin-LF | Schedule 1 Dose Escalation Cohort: 1.5 mg/m^2 Eribulin-LF | Schedule 2 Dose Escalation Cohort: 1.0 mg/m^2 Eribulin-LF | Schedule 2 Dose Escalation Cohort: 1.5 mg/m^2 Eribulin-LF | Schedule 2 Dose Escalation Cohort: 2.0 mg/m^2 Eribulin-LF
Number analyzed (Participants) | 6 | 6 | 7 | 3 | 9 | 3
mL | 1953.3 (547.53) | 2091.7 (505.03) | 2310.0 (514.39) | 3793.3 (1866.61) | 2873.3 (1530.20) | 1993.3 (96.09)

11. Secondary Outcome: Renal Clearance (CLr) of Eribulin-LF
Description: Blood samples for Schedule 1 were drawn on Cycle 1/Day 1 and Cycle 3/Day 1 predose, 15 min after SOI, 5 min after EOI, 0.5, 1, 2, 4, 6, 8, and 24 h postdose, and Day 4, Day 7, Day 9, and Day 11. Blood samples for Schedule 2 were drawn on Cycle 1/Day 1 and Day 15 and Cycle 3/Day 1 and Day 15 predose, 15 min after SOI, 5 min after EOI, 0.5, 1, 2, 4, 6, 8, and 24 h postdose, and Day 4, Day 7, Day 9 and Day 11. Some participants followed a different PK assessment schedule prior to protocol amendment 3. Plasma concentrations of eribulin-LF were determined using a validated LC/MS/MS method. Plasma PK data were analyzed using a noncompartmental analysis approach to obtain individual participant estimates of CLr, which was then summarized as the mean and standard deviation for all participants and expressed in liters/hour (L/hr).
Time Frame: Schedule 1: Cycle 1/Day 1 and Cycle 3/Day 1; Schedule 2: Cycle 1/Day 1 and Day 15 and Cycle 3/Day 1 and Day 15
Population: The PK analysis set was the group of participants who had sufficient PK data to derive at least one PK parameter.
Measure: Mean (Standard Deviation); unit: mL/h
Arm/Group | Schedule 1 Dose Escalation Cohort: 1.0 mg/m^2 Eribulin-LF | Schedule 1 Dose Escalation Cohort: 1.4 mg/m^2 Eribulin-LF | Schedule 1 Dose Escalation Cohort: 1.5 mg/m^2 Eribulin-LF | Schedule 2 Dose Escalation Cohort: 1.0 mg/m^2 Eribulin-LF | Schedule 2 Dose Escalation Cohort: 1.5 mg/m^2 Eribulin-LF | Schedule 2 Dose Escalation Cohort: 2.0 mg/m^2 Eribulin-LF
Number analyzed (Participants) | 4 | 5 | 5 | 1 | 5 | 3
mL/h | 4.833 (1.8621) | 8.698 (3.6476) | 13.316 (12.7962) | 3.800 | 5.957 (5.8697) | 4.843 (0.9514)

12. Secondary Outcome: Fraction of Unchanged Eribulin-LF Excreted in the Urine (fe)
Description: Urinalysis was performed at Screening, Baseline, Cycle 1/Day 15, and each study visit of every cycle thereafter. If urinalysis suggested a urinary tract infection, or if clinically indicated, a urine microscopy, culture, and sensitivity was to be performed at the institution's laboratory. If urine protein was ≥ 2+ on urinalysis, then a 24-hour urine collection was to be done to quantify the 24-hour urine protein excretion. The samples were analyzed for the amount of eribulin in the urine using liquid LC/MS method of analysis. Urine PK data were analyzed using a noncompartmental analysis approach to obtain individual participant estimates of fe, which was then summarized as the mean and standard deviation for all participants and expressed in percentage of eribulin-LF.
Time Frame: Schedule 1: Cycle 1/Day 1 and Cycle 3/Day 1; Schedule 2: Cycle 1/Day 1 and Day 15 and Cycle 3/Day 1 and Day 15
Population: The PK analysis set was the group of participants who had sufficient PK data to derive at least one PK parameter.
Measure: Mean (Standard Deviation); unit: percent of eribulin-LF
Arm/Group | Schedule 1 Dose Escalation Cohort: 1.0 mg/m^2 Eribulin-LF | Schedule 1 Dose Escalation Cohort: 1.4 mg/m^2 Eribulin-LF | Schedule 1 Dose Escalation Cohort: 1.5 mg/m^2 Eribulin-LF | Schedule 2 Dose Escalation Cohort: 1.0 mg/m^2 Eribulin-LF | Schedule 2 Dose Escalation Cohort: 1.5 mg/m^2 Eribulin-LF | Schedule 2 Dose Escalation Cohort: 2.0 mg/m^2 Eribulin-LF
Number analyzed (Participants) | 4 | 5 | 5 | 1 | 5 | 3
percent of eribulin-LF | 7.28 (1.597) | 9.88 (2.558) | 13.78 (7.379) | 4.70 | 6.56 (5.327) | 7.30 (2.254)

13. Secondary Outcome: Percentage of Participants With Best Overall Response (BOR)
Description: BOR to treatment was assessed according to Response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.1. BOR was the best confirmed response of complete response (CR), partial response (PR), progressive disease (PD), stable disease (SD), or not evaluable (NE), recorded from the start of eribulin-LF until disease progression/recurrence or death. CR; disappearance of all target lesions for at least 1 month. PR; at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. PD; at least 20% or greater increase in the sum of the longest diameter of measured lesions, taking as reference the smallest sum of the longest diameter recorded since treatment started or the appearance of one or more new lesions. SD; PR failed to be achieved in the overall response assessment and there was no PD observed at the end of 6 cycles or later after starting eribulin-LF.
Time Frame: Baseline to first date of documented CR, PR, SD, or PD, assessed up to data cutoff date (17 May 2016), for up to approximately 3 years 7 months
Population: The SAS was the group of participants who received study drug and had at least 1 post-dose safety assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Schedule 1 Dose Escalation Cohort: 1.0 mg/m^2 Eribulin-LF | Schedule 1 Dose Escalation Cohort: 1.4 mg/m^2 Eribulin-LF | Schedule 1 Dose Escalation Cohort: 1.5 mg/m^2 Eribulin-LF | Schedule 2 Dose Escalation Cohort: 1.0 mg/m^2 Eribulin-LF | Schedule 2 Dose Escalation Cohort: 1.5 mg/m^2 Eribulin-LF | Schedule 2 Dose Escalation Cohort: 2.0 mg/m^2 Eribulin-LF | Schedule 2 Expansion Cohort: 1.5 mg/m^2 Eribulin-LF
Number analyzed (Participants) | 7 | 6 | 7 | 3 | 9 | 3 | 23
percentage of participants
  CR | 0 | 0 | 0 | 0 | 0 | 0 | 0
  PR | 14.3 | 16.7 | 0 | 0 | 0 | 33.3 | 13.0
  SD | 71.4 | 16.7 | 57.1 | 33.3 | 11.1 | 0 | 34.8
  PD | 0 | 66.7 | 42.9 | 33.3 | 66.7 | 66.7 | 43.5
  Unknown | 14.3 | 0 | 0 | 33.3 | 22.2 | 0 | 8.7

14. Secondary Outcome: Percentage of Participants With Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants with BOR of CR or PR based on RECIST v1.1 criteria or target lesions assessed by magnetic resonance imaging/computed tomography (MRI/CT) scans, as determined by independent radiologic review. BOR of CR was confirmed by a subsequent CR assessment at least 4 weeks later. BOR of PR was confirmed by a subsequent CR or PR assessment at least 4 weeks later. CR was defined as disappearance of all target lesions. Any pathological lymph nodes (target or non-target) had to be reduced in short axis to less than 10 mm. PR was defined as at least a 30% decrease in sum of diameters of target lesions, taking as reference the baseline sum of diameters. The null hypothesis ORR was less than or equal to 10% was tested using 1-sided exact test of a single proportion, at 1-sided 0.05 level. ORR was presented with corresponding 2-sided, 95% confidence interval (CI). ORR=CR+PR.
Time Frame: From date of treatment start until disease progression, development of unacceptable toxicity, withdrawal of consent, participant's choice to stop study treatment, or up to data cutoff date (17 May 2016), for up to approximately 3 years 7 months
Population: The SAS was the group of participants who received study drug and had at least 1 post-dose safety assessment.
Measure: Median (95% Confidence Interval); unit: percentage of participants
Arm/Group | Schedule 1 Dose Escalation Cohort: 1.0 mg/m^2 Eribulin-LF | Schedule 1 Dose Escalation Cohort: 1.4 mg/m^2 Eribulin-LF | Schedule 1 Dose Escalation Cohort: 1.5 mg/m^2 Eribulin-LF | Schedule 2 Dose Escalation Cohort: 1.0 mg/m^2 Eribulin-LF | Schedule 2 Dose Escalation Cohort: 1.5 mg/m^2 Eribulin-LF | Schedule 2 Dose Escalation Cohort: 2.0 mg/m^2 Eribulin-LF | Schedule 2 Expansion Cohort: 1.5 mg/m^2 Eribulin-LF
Number analyzed (Participants) | 7 | 6 | 7 | 3 | 9 | 3 | 23
percentage of participants | 14.3 [0.4 to 57.9] | 16.7 [0.4 to 64.1] | 0 [0.0 to 41.0] | 0 [0.0 to 70.8] | 0 [0.0 to 33.6] | 33.3 [0.8 to 90.6] | 13.0 [2.8 to 33.6]

15. Secondary Outcome: Percentage of Participants With Disease Control Rate (DCR)
Description: DCR was the percentage of the participants who had BOR of CR, PR, and SD, based on assessments by each site investigator using RECIST v1.1. The minimum duration of SD was defined as 5 weeks (or 7 weeks for Schedules 1a and 2 in the Dose Escalation Part) following the date of the first dose of study drug in order for stable disease to be considered the best overall response. The 95% CI was constructed using the method of Clopper and Pearson. DCR = CR + PR + SD
Time Frame: as for outcome 14
Population: The SAS was the group of participants who received study drug and had at least 1 post-dose safety assessment.
Measure: Median (95% Confidence Interval); unit: percentage of participants
Arm/Group | Schedule 1 Dose Escalation Cohort: 1.0 mg/m^2 Eribulin-LF | Schedule 1 Dose Escalation Cohort: 1.4 mg/m^2 Eribulin-LF | Schedule 1 Dose Escalation Cohort: 1.5 mg/m^2 Eribulin-LF | Schedule 2 Dose Escalation Cohort: 1.0 mg/m^2 Eribulin-LF | Schedule 2 Dose Escalation Cohort: 1.5 mg/m^2 Eribulin-LF | Schedule 2 Dose Escalation Cohort: 2.0 mg/m^2 Eribulin-LF | Schedule 2 Expansion Cohort: 1.5 mg/m^2 Eribulin-LF
Number analyzed (Participants) | 7 | 6 | 7 | 3 | 9 | 3 | 23
percentage of participants | 85.7 [42.1 to 99.6] | 33.3 [4.3 to 77.7] | 57.1 [18.4 to 90.1] | 33.3 [0.8 to 90.6] | 11.1 [0.3 to 48.2] | 33.3 [0.8 to 90.6] | 47.8 [26.8 to 69.4]

16. Secondary Outcome: Percentage of Participants With Clinical Benefit Rate (CBR)
Description: CBR was defined as the percentage of participants with BOR of CR or PR or durable stable disease (dSD) [CR + PR + dSD] based on RECIST v1.1. The dSD rate was defined as the percentage of participants with dSD (based on RECIST 1.1 and defined as SD lasting greater than or equal to 6 months), as determined by the site Investigator.
Time Frame: as for outcome 14
Population: The SAS was the group of participants who received study drug and had at least 1 post-dose safety assessment.
Measure: Median (95% Confidence Interval); unit: percentage of participants
Arm/Group | Schedule 1 Dose Escalation Cohort: 1.0 mg/m^2 Eribulin-LF | Schedule 1 Dose Escalation Cohort: 1.4 mg/m^2 Eribulin-LF | Schedule 1 Dose Escalation Cohort: 1.5 mg/m^2 Eribulin-LF | Schedule 2 Dose Escalation Cohort: 1.0 mg/m^2 Eribulin-LF | Schedule 2 Dose Escalation Cohort: 1.5 mg/m^2 Eribulin-LF | Schedule 2 Dose Escalation Cohort: 2.0 mg/m^2 Eribulin-LF | Schedule 2 Expansion Cohort: 1.5 mg/m^2 Eribulin-LF
Number analyzed (Participants) | 7 | 6 | 7 | 3 | 9 | 3 | 23
percentage of participants | 28.6 [3.7 to 71.0] | 33.3 [4.3 to 77.7] | 0 [0.0 to 41.0] | 0 [0.0 to 70.8] | 0 [0.0 to 33.6] | 33.3 [0.8 to 90.6] | 17.4 [5.0 to 38.8]

17. Secondary Outcome: Percentage of Participants With Progression Free Survival (PFS)
Description: PFS was defined as the time from the date of treatment start until progressive disease or death from any cause in the absence of progressive disease. Disease progression was defined as at least a 20% increase in the sum of the longest diameter of target lesions (taking as reference the smallest sum on study), recorded since the treatment started or the appearance of 1 or more new lesions as assessed by IRR using RECIST v1.1. The duration of PFS was calculated as end date minus date of first drug plus 1, based on assessments by the site Investigator. PFS was calculated using Kaplan-Meier estimate and presented with 2-sided 95% Cl.
Time Frame: as for outcome 14
Population: PFS data was not collected as this is a Phase I dose escalation design and was not the focus of the study.
Arm/Group | Schedule 1: Total Escalation Cohorts | Schedule 2: Total Dose Escalation and Expansion
Number analyzed (Participants) | 0 | 0

18. Secondary Outcome: Number of Participants With the Indicated Shift From Baseline Category to the Indicated Worst Post-Baseline Category
Description: The effects of eribulin-LF on cardiovascular repolarization were evaluated via 24-hour, 12-lead continuous Holter electrocardiogram (ECG) monitoring in Cycle 1, Day 1 for Schedule 1 and Day 1 and Day 15 of Schedule 2. Individual ECGs were extracted in triplicate from the Holter recordings at specified time points and were evaluated by a central laboratory. QT intervals were measured from Lead II and were corrected for heart rate (QTc) using Fridericia's (QTcF) and Bazett's (QTcB) correction factors. The primary QTc parameter was QTcF. Secondary parameters (QTcB, QT, QRS, and hazard ratio/heart rate (HR)) and waveforms (T-waves) were evaluated. BL= Baseline, PBL = post-Baseline, A,NCS = abnormal, not clinically significant, A, CS = abnormal, clinically significant
Time Frame: Baseline (Day -1), Schedule 1 (Cycle 1 Day 1); Schedule 2 (Cycle 1 Day 1 and Day 15)
Population: The SAS was the group of participants who received study drug and had at least 1 post-dose safety assessment. Only participants with baseline and post-baseline values were reported.
Measure: Count of Participants; unit: Participants
Arm/Group | Schedule 1 Dose Escalation Cohort: 1.0 mg/m^2 Eribulin-LF | Schedule 1 Dose Escalation Cohort: 1.4 mg/m^2 Eribulin-LF | Schedule 1 Dose Escalation Cohort: 1.5 mg/m^2 Eribulin-LF | Schedule 2 Dose Escalation Cohort: 1.0 mg/m^2 Eribulin-LF | Schedule 2 Dose Escalation Cohort: 1.5 mg/m^2 Eribulin-LF | Schedule 2 Dose Escalation Cohort: 2.0 mg/m^2 Eribulin-LF | Schedule 2 Expansion Cohort: 1.5 mg/m^2 Eribulin-LF
Number analyzed (Participants) | 7 | 6 | 7 | 3 | 9 | 3 | 23
Participants
  BL=normal to PBL=normal | 3 | 4 | 6 | 2 | 4 | 2 | 14
  BL=normal to PBL=A,NCS | 0 | 0 | 0 | 0 | 0 | 0 | 0
  BL=normal to PBL=A,CS | 3 | 0 | 0 | 0 | 2 | 0 | 5
  BL=A,NCS to PBL=normal | 0 | 0 | 0 | 0 | 0 | 0 | 0
  BL=A,NCS to PBL=A,NCS | 0 | 0 | 0 | 0 | 0 | 0 | 0
  BL=A,NCS to PBL=A,CS | 0 | 0 | 0 | 0 | 0 | 0 | 0
  BL=A,CS to PBL=normal | 0 | 0 | 0 | 0 | 0 | 0 | 1
  BL=A,CS to PBL=A,NCS | 0 | 0 | 0 | 0 | 0 | 0 | 0
  BL=A,CS to PBL=A,CS | 1 | 2 | 1 | 1 | 2 | 1 | 3

ADVERSE EVENTS:
Time Frame: From date of first dose until 30 days after the final dose of study drug, up to approximately 3 years 8 months
Description: Treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs) were reported for the Safety Analysis Set. All adverse events were graded using Common Terminology Criteria for Adverse Events (CTCAE) version 4.1. Participants who did not receive treatment were not analyzed.
Arm/Group | Schedule 1 Dose Escalation Cohort: 1.0 mg/m^2 Eribulin-LF | Schedule 1 Dose Escalation Cohort: 1.4 mg/m^2 Eribulin-LF | Schedule 1 Dose Escalation Cohort: 1.5 mg/m^2 Eribulin-LF | Schedule 2 Dose Escalation Cohort: 1.0 mg/m^2 Eribulin-LF | Schedule 2 Dose Escalation Cohort: 1.5 mg/m^2 Eribulin-LF | Schedule 2 Dose Escalation Cohort: 2.0 mg/m^2 Eribulin-LF | Schedule 2 Expansion Cohort: 1.5 mg/m^2 Eribulin-LF
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/6 | 0/7 | 0/3 | 0/9 | 0/3 | 0/23
Serious Adverse Events (participants affected / at risk) | 1/7 | 2/6 | 6/7 | 1/3 | 3/9 | 2/3 | 9/23
Other Adverse Events (participants affected / at risk) | 7/7 | 6/6 | 7/7 | 3/3 | 8/9 | 3/3 | 23/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Schedule 1 Dose Escalation Cohort: 1.0 mg/m^2 Eribulin-LF (N=7) | Schedule 1 Dose Escalation Cohort: 1.4 mg/m^2 Eribulin-LF (N=6) | Schedule 1 Dose Escalation Cohort: 1.5 mg/m^2 Eribulin-LF (N=7) | Schedule 2 Dose Escalation Cohort: 1.0 mg/m^2 Eribulin-LF (N=3) | Schedule 2 Dose Escalation Cohort: 1.5 mg/m^2 Eribulin-LF (N=9) | Schedule 2 Dose Escalation Cohort: 2.0 mg/m^2 Eribulin-LF (N=3) | Schedule 2 Expansion Cohort: 1.5 mg/m^2 Eribulin-LF (N=23)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 2
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Device leakage (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Device occlusion (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 1 | 2 | 0 | 2 | 0 | 2
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neutropenic sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Transaminases increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Spinal cord compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Schedule 1 Dose Escalation Cohort: 1.0 mg/m^2 Eribulin-LF (N=7) | Schedule 1 Dose Escalation Cohort: 1.4 mg/m^2 Eribulin-LF (N=6) | Schedule 1 Dose Escalation Cohort: 1.5 mg/m^2 Eribulin-LF (N=7) | Schedule 2 Dose Escalation Cohort: 1.0 mg/m^2 Eribulin-LF (N=3) | Schedule 2 Dose Escalation Cohort: 1.5 mg/m^2 Eribulin-LF (N=9) | Schedule 2 Dose Escalation Cohort: 2.0 mg/m^2 Eribulin-LF (N=3) | Schedule 2 Expansion Cohort: 1.5 mg/m^2 Eribulin-LF (N=23)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 2
Neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 1 | 0 | 1 | 3 | 10
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cushingoid (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 2
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 1 | 2 | 0 | 0 | 3
Diarrhoea (Gastrointestinal disorders) | 5 | 1 | 2 | 1 | 3 | 0 | 4
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 2 | 1 | 4
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 5
Constipation (Gastrointestinal disorders) | 2 | 3 | 3 | 0 | 0 | 0 | 6
Nausea (Gastrointestinal disorders) | 3 | 1 | 1 | 1 | 2 | 1 | 11
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Lip disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lip dry (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oesophageal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Paraesthesia oral (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 3
Fatigue (General disorders) | 2 | 3 | 2 | 0 | 2 | 1 | 9
Face oedema (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Infusion site erythema (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Suprapubic pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hepatitis fulminant (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 2
Oral candidiasis (Infections and infestations) | 2 | 2 | 1 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 3 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 2
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 4
Gastrointestinal bacterial infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Viral rhinitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 | 1
Weight decreased (Investigations) | 0 | 1 | 1 | 1 | 0 | 1 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood magnesium decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood magnesium increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood uric acid increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 4 | 2 | 4 | 1 | 1 | 0 | 5
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 3
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 2 | 1 | 0 | 0 | 0 | 1
Lethargy (Nervous system disorders) | 4 | 0 | 1 | 2 | 1 | 2 | 3
Headache (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 4
Neurotoxicity (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1
Chromaturia (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vulvovaginal pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 0 | 1 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 3 | 4 | 1 | 2 | 2 | 8
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin mass (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Spider naevus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Hot flush (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vasodilatation (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other